CLINICAL TRIAL: NCT05803031
Title: Efficacy of Locally Delivered Tea Tree Oil Gel as an Adjunct to Non-Surgical Periodontal Management (A Randomized Controlled Clinical Trial With Biochemical Analysis)
Brief Title: Efficacy of Locally Delivered Tea Tree Oil Gel as an Adjunct to Non-Surgical Periodontal Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1045
Record Dates: First submitted 2023-02-12; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Periodontal Pocket
Keywords: Local Drug Delivery; Periodontitis; Tea Tree Oil
MeSH Terms: conditions — Periodontal Pocket; Periodontitis | interventions — Tea Tree Oil

STUDY DESIGN:
Intervention Model Description: This study was designed to be a Randomized, Controlled, Parallel design, Two arms clinical trial. The patients will be randomly allocated to one of the two groups; test and control group using computer generated random tables (www.randomizer.org ) .
Who Masked: Participant
Masking Description: Patients will be blinded to the type of the intervention and the whole-time frame of the study will be 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Test group) (Experimental): Eleven patients with localized periodontitis, receiving full mouth non-surgical periodontal debridement followed by local delivery of tea tree oil gel as an adjunctive treatment.
  Interventions: Drug: Melaleuca Alternifolia Oil; Procedure: Non-surgical periodontal debridement
- Group II (Control group) (Placebo Comparator): Eleven patients with localized periodontitis, receiving full mouth non-surgical periodontal debridement only.
  Interventions: Procedure: Non-surgical periodontal debridement

INTERVENTIONS:
Drug: Melaleuca Alternifolia Oil — Tea tree oil 5% gel (Sigma Aldrich® Steinheim, Germany) for local sub gingival application was prepared by the Department of Pharmaceutics, Faculty of Pharmacy.
  The gelling agent; Carbopol 940 (1% w/v) was first soaked in distilled water for 2 h then TTO dissolved in an appropriate amount of propylene glycol was added to the Carbopol dispersion. Methyl paraben 0.2% w/v dissolved in preheated water was used as a preservative. The gel mixture was then magnetically stirred for 30 min. Finally, pH was adjusted using 1 N NaOH added dropwise with gentle stirring with a spatula until the desired pH value (6.5-7) was reached. The gel was sterilized by autoclaving at 110 °C for 20 min.
  Arms: Group I (Test group)
Procedure: Non-surgical periodontal debridement — Scaling and root surface debridement

SUMMARY:
Periodontitis is an inflammatory disease of the teeth's supporting tissues caused by specific microbes or groups of microorganisms that contributes to gradual deterioration of the periodontal ligament and alveolar bone, leading to periodontal pockets, gingival recession, or both. Periodontitis is generally known to be caused by the continuous destruction of the surrounding periodontium by complexly organized bacterial communities that colonizes the tooth surface, gingival margin, and subgingival area in the form of dental plaque biofilm. Researchers suggest the dependence of the treatment of periodontal disease on controlling the residual mass of periodontal microbes. Therefore, it is proposed that non-surgical therapy is regarded as the initial treatment of periodontitis, which includes mechanical therapy, such as oral hygiene measures and mechanical debridement like scaling and root planning. Chemical therapy could supplement the non-surgical mechanical therapy, including antimicrobials that can be systemically or locally delivered. Systemic delivery of antimicrobials plays a critical role in reaching microorganisms dispersed in the oral cavity, including those in non-dental oral niches, such as the dorsum of the tongue and crypts of tonsils. Despite these advantages, it might lead to unwanted systemic effects -such as nausea, vomiting, and gastrointestinal discomfort- or bacterial resistance, as it is completely dependent on the patient's adherence. Local Drug Delivery (LDD), compared to systemic administration, provides higher therapeutic concentrations of antibiotics at site of infection that is inaccessible to the systemic route and it is independent of patient's adherence, as has been shown in various studies. Natural products have long been an important source of medications, with natural ingredients accounting for almost half of all pharmaceuticals currently in use. Oriental medicines have been studied for their antibacterial and anti-inflammatory properties, as well as periodontal tissue regeneration, in the treatment of periodontal disease. Tea tree oil (TTO), which is an example of one of these natural products, is obtained from paper bark tea tree. Tea tree oil was made from natural bush stands of plants, allegedly Melaleuca alternifolia, that generated oil with the required chemotype during that early stage. Melaleuca alternifolia's native habitat is low-lying, swampy, subtropical coastal ground along the Clarence and Richmond Rivers in northeastern New South Wales and southern Queensland, and it does not occur natively beyond Australia, unlike numerous other Melaleuca species. Tea tree oil, commonly known as "oil of the Tea tree" or "Melaleuca essential oil," is one of the most well-known essential oils. It's made from the Melaleuca alternifolia tree's leaves, which have been distilled. This plant is a member of the Myrtaceae family, which includes Australian arboreal plants. It is known as "nature's most versatile healer" among the native populations. Tea tree oil (TTO) possesses antibacterial, anti-inflammatory, antifungal, antiviral, antioxidant, and antiprotozoal properties. Components of tea tree oil include: Terpinen-4-ol, α-Terpinene, γ -Terpinene, 1,8-Cineole, α -Terpinolene, p-Cymene, (+)-α-Pinene, α -Terpineol, Aromadendrene, δ -Cadinene, (+)-Limonene, Sabinene, and Globulol. The capacity of TTO components to reduce the production of TNF α, IL-1beta, IL-8, IL-10, and PGE2 by lipopolysaccharide activated human monocytes shows TTO's anti-inflammatory action, according to the researchers. TTO's major active components are 1,8-cineole and Terpinen-4-ol, and it has been shown that 1,8-cineole possesses anti-inflammatory characteristics and may permeate human skin. Other research suggests that Terpinen-4-ol not only has anti-inflammatory characteristics like 1,8-cineol, but also has anti-bacterial capabilities. TTO has the same antibacterial effect as chlorhexidine (CHX), however the mode of action is different. Antibacterial, antiviral, and antifungal activities are all present. According to researches, TTO is capable of lowering both inflammatory mediators and periodontal pathogens, which in turn reduces the stimulation of inflammatory cytokines, allowing periodontal tissues to repair when applied locally in periodontal pockets. Melaleuca Alternifolia was chosen for this study as a local drug delivery in the gel form to be placed in periodontal pockets as an adjunct to non-surgical periodontal debridement for the management of localized periodontitis due to its therapeutic effects, ease of availability of tea tree oil, cost effectiveness, and safety with no adverse reactions.

DETAILED DESCRIPTION:
Aim & objectives of the Study:

The aim of this randomized controlled clinical and biochemical trial is to assess the efficacy of locally applied Melaleuca Alternifolia (tea tree oil) gel as a supplement to non-surgical periodontal debridement in the treatment of patients with localized periodontitis.

Primary objectives:

* Assess the effectiveness of tea tree oil gel in the management of periodontitis using clinical parameters.
* Evaluate Patients' satisfaction using the patient satisfaction questionnaire.

Secondary objective:

• Determine the impact of tea tree oil gel on the level of Tumor Necrosis Factor (TNF-α) in the gingival crevicular fluid.

Treatment protocol and intervention:

* Preoperative periapical radiographs will be done initially to determine the level of bone using a standard periapical parallel technique with digital sensor.
* The patients will undergo full mouth one stage debridement using ultrasonic scalers, manual scalers and curettes.
* Full mouth periodontal charting and samples from gingival crevicular fluid will be obtained using a sterile perio-paper inserted into the deepest periodontal pocket with horizontal bone loss immediately after finishing phase I therapy.
* Melaleuca Alternifolia Gel will be gently administered in the deepest pocket by syringe with blunt tip and the syringe will be removed slowly to avoid injuring the tissues for group I patients after phase 1 therapy by two weeks.
* After 3 months of phase I therapy, the patients will be followed up with evaluation of the clinical parameters.

Social & scientific values: Provide the dentists a more convenient way to reduce periodontal pockets in periodontitis patient by locally applying Melaleuca Alternifolia gel as an adjunct to non-surgical periodontal debridement.

Risks to study participants: The participants are not subjected to any risks.

Benefits to study participants:

Since the main objective of the research is using tea tree oil as a local delivery drug in the gel form to be placed in periodontal pockets as an adjunct to non-surgical periodontal debridement for the management of localized periodontitis, the benefit of the research is to provide the patient better therapeutic effect and a safe local delivery drug with no adverse reactions.

Benefits of the study to the community: Determination of the impact of tea tree oil gel on the level of Tumor necrosis factor-alpha (TNF-α) in the gingival crevicular fluid.

Privacy, Record keeping & confidentiality: All patients' data, information and study results will be kept under strict confidentiality and will be stored and kept as required. Only the primary researcher and the main investigator will have access to such data during the period of the study. At the end of the study all participants will be informed with the results and outcomes of the study as well as any health issues if found concerning them.

The study has been approved and accepted by the Diagnosis, Oral Medicine and Periodontology Department as approved by the endorsement released from the departments' committee with the code: OMD-2021-11 on Sunday 7/11/2020.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with age range of 25-50years.
2. Patients diagnosed to have (Stage II or Stage III) periodontitis; (3-6 mm CAL, pocket depth ≤ 7 mm, mostly horizontal 15%-33% bone loss as assessed by preoperative radiographs with no tooth loss due to periodontitis).
3. Systemic (medically) free patients.
4. Patients who can follow and maintain oral hygiene instructions.

Exclusion Criteria:

1. Pregnant ladies or lactating mothers.
2. Smokers.
3. Patients with history of allergy against one of the components of tea tree oil.
4. Asthmatic patients.
5. Periodontal therapy in the last 6 months

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Probing Depth | 3 months
  Measured in mm from gingival margin to periodontal pocket using a periodontal probe.
Evaluate Patients' satisfaction | 3 months
  The response choices requested the patients to assign a 5-point rating scale to each item. Responses would be rated from 1 to 5, with 1 being a total disagree and 5 representing a total agreement. Higher scores therefore represent better patient satisfaction.
Clinical attachment level | 3 months
  Measured in mm from cemento-enamel junction to the depth of the periodontal pocket.

SECONDARY OUTCOMES:
Level of Tumor Necrosis Factor (TNF-α) in the gingival crevicular fluid | 3 months
  GCF will be collected with sterile periopaper strips. The periopaper should be gently inserted into the gingival crevice until slight resistance is felt.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt